CLINICAL TRIAL: NCT05508646
Title: Group-Based Telehealth Music Therapy Intervention for Patients With Dementia: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0409
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia
MeSH Terms: conditions — Behavior; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Twelve participants will be randomized for the intervention. The music therapy intervention takes place once a week for 6 weeks via telemedicine, with the first session reserved for music therapy intake/assessment. There are 5 additional visits, once per week. The format of the sessions may include: a greeting song to orient the participant to the start of the session; singing of 1-3 preferred/chosen songs to address cognition and communication; two movement songs with instrument playing interventions to stimulate cognition and movement; songwriting for self-expression, cognitive, and emotional support; relaxation/mindfulness; a closing song to help the participant transition at the completion of the session, The music therapist also provides training to caregivers in techniques to utilize music for behavioral support.
  Interventions: Behavioral: Music therapy intervention
- Control arm (Other): Twelve participants will be randomized to receive a personalized music CD that they keep and can listen to as they wish.
  Interventions: Behavioral: Personalized music CD

INTERVENTIONS:
Behavioral: Music therapy intervention — The format of the sessions may include: a greeting song to orient the participant to the start of the session; singing of 1-3 preferred/chosen songs to address cognition and communication; two movement songs with instrument playing interventions to stimulate cognition and movement; songwriting for self-expression, cognitive, and emotional support; relaxation/mindfulness; a closing song to help the participant transition at the completion of the session, The music therapist also provides training to caregivers in techniques to utilize music for behavioral support.
  Arms: Intervention arm
Behavioral: Personalized music CD — Participants will receive a personalized music CD that they keep and can listen to as they wish.
  Arms: Control arm

SUMMARY:
Twelve participants and their care partners will be randomized for the intervention. The music therapy intervention takes place once a week for 6 weeks via telemedicine, with the first session reserved for music therapy intake/assessment. There are 5 additional visits, once per week. The format of the sessions may include: a greeting song to orient the participant to the start of the session; singing of 1-3 preferred/chosen songs to address cognition and communication; two movement songs with instrument playing interventions to stimulate cognition and movement; songwriting for self-expression, cognitive, and emotional support; relaxation/mindfulness; a closing song to help the participant transition at the completion of the session, The music therapist also provides training to caregivers in techniques to utilize music for behavioral support.

Twelve participants and their care partners will be randomized to receive a personalized music CD that they keep and can listen to as they wish.

DETAILED DESCRIPTION:
This is a single-blinded prospective randomized control pilot study. We are aiming to recruit 24 participants, with their caregiver, who have mild to moderate dementia from Geisinger Memory and Cognition Program. 12 participants will be randomized for the music intervention arm, and 12 for the control arm. The music therapy intervention takes place once a week for 6 weeks via telemedicine. 12 participants will be randomized to receive a music CD with a personalized playlist. At baseline and end of study several measures will be completed: Mini-mental State Examination and the Geriatric Depression Scale by the participant; and the caregiver will complete the Neuropsychiatric Inventory-Severity/Distress scales, Modified Caregiver Stain Index and Patient Health Questionnaire-9 at those times as well as at 6 weeks. The music therapist will fill out an engagement form for each session she has with the participant. The primary outcome is to compare pre- and post-scores on measures of cognition, BPSD, caregiver strain, and depression for participant and caregiver for those undergoing the telehealth music therapy intervention vs. those who receive a personalized music selection on CD. We also aim to explore whether degree of engagement during music therapy affects outcomes in Aim 1.

With significant economic and emotional impacts, caregiving for patients with dementia is stressful. BPSD associated with dementia leads to increased stress for people with dementia and their loved ones and may lead to earlier nursing home placement. If behavioral symptoms of persons with dementia could be alleviated, caregivers may feel more empowered, and patients with dementia may be able to stay at home longer. Music therapy has been shown to help with behaviors, agitation, and depression, and may help decrease caregiver stress. We are hoping through this study to show that using a telehealth platform, music therapy is feasible for patients who would not otherwise have access to it.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for participants:

* Mild to moderate dementia (MMSE 13-26 at their last clinic visit, if within 6 months)
* English-speaking
* Auditory acuity adequate for participating with music therapy
* Access to high-speed internet, webcam, and a microphone
* A caregiver willing to participate

Inclusion Criteria for Caregivers:

* Must be an adult relative, friend, or caretaker (non-professional)
* English speaking
* Visual and auditory acuity adequate for communicating with examiner and completing questionnaires

Exclusion Criteria:

Exclusion Criteria for participants:

* Must not be presently participating in another interventional study
* Must not demonstrate increased anxiety/distress when utilizing a telehealth platform
* Must not have received a clinical prognosis of rapidly progressing dementia

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination | 1 year
  The Mini Mental State Examination is a 30-point questionnaire used to measure cognitive impairment. Any score of 24 or more indicates a normal cognition. Scores of ≤9 points can indicate severe, 10-18 points moderate or 19-23 points mild cognitive impairment.
Geriatric Depression Scale | 1 year
  The Geriatric Depression Scale is a 30-item questionnaire used to measure depression in older populations. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Neuropsychiatric Inventory-Severity/Distress scales | 1 year
  The Neuropsychiatric Inventory-Severity/Distress scales are used to determine the severity of the participants' neuropsychiatric symptoms and the distress these cause the caregiver. The severity scale has scores ranging from 1 to 3 points (1=mild; 2=moderate; and 3=severe) and the scale for assessing caregiver distress has scores ranging from 0 to 5 points (0=no distress; 1=minimal distress; 2=mild distress; 3=moderate distress; 4=severe distress; and 5=extreme distress).
Modified Caregiver Strain Index | 1 year
  The Modified Caregiver Strain Index uses 13 questions to measure strain related to caregiving. Scoring ranges from 26 to 0. Each 'yes' equals 2 points, each 'sometimes' equals 1 point, and each 'no' equals 0 points. A higher score indicates a higher level of caregiver strain.
Patient Health Questionnaire-9 | 1 year
  Patient Health Questionnaire-9 uses 9 questions to measure the caregivers' symptoms of depression. Scoring ranges from 27 to 0. Scores ranging from 0 to 4 points are considered normal/minimal. Scores ranging from 5 to 9 points are considered mild depression severity. Scores ranging from 10 to 14 points are considered moderate depression severity. Scores ranging from 15 to 19 points are considered moderately severe depression severity. Scores ranging from 20 to 27 points are considered severe depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Lichtenstein, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Maya Lichtenstein, Wilkes-Barre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No